CLINICAL TRIAL: NCT03671668
Title: Crestal Bone Loss and Patient Satisfaction of Screw Retained Restoration Using Multi-unit Abutments Versus Intra-oral Luting on Titanium Bases in Implant Supported Complete Overdentures: A Randomized Clinical Trial
Brief Title: Crestal Bone Loss and Patient Satisfaction of Screw Retained Restoration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed saber mohamed ahmed, Assistant lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28905011809519
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Completely edentulous patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screw retained prosthesis on transmucosal abutments (Active Comparator)
  Interventions: Other: titanium bases using intra oral luting cement technique
- Screw retained prosthesis on titanium bases (Experimental)
  Interventions: Other: titanium bases using intra oral luting cement technique

INTERVENTIONS:
Other: titanium bases using intra oral luting cement technique — comparing between screw retained prosthesis constructed on transmucosal abutments versus titanium bases in terms of crestal bone loss and patient satisfaction

SUMMARY:
On of the main fixed prosthetic options of completely edentulous patients is the screw-retained implant supported prosthesis which was constructed on transmucosal abutments with its encountered problems such as: hardness to make it passively seated with multiple screw fracture and loosening problems and multiple encountered veneer material fracture and so there effect on patient satisfaction with multiple maintenance recalls.so, we want to try a new technique of fabrication which was proposed for reducing the problems of lack of passivity which is the intraoral luting cement technique on titanium bases with reduced screw number but, with luting cement problems as de-cementation and cement biological effects on soft tissues and bone and there effect on number of patient recall visits and maintenance and so there effect on patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients
* Patients with completely edentulous ridges have an opposing natural dentition or implant supported overdenture
* Completely edentulous patients (with the above mentioned criteria) who have proper amount of attached gingiva (≥2 mm) or to be created
* Completely edentulous patients (with the above mentioned criteria) who have no history of bruxism
* Completely edentulous patients (with the above mentioned criteria) who were free or controlled diabetic assessed by measuring glycosylated haemoglobin (HbA1c). (lesser than or equal to 6.4 percent )

Exclusion Criteria:

* Patients having a medical condition that absolutely contraindicates implant placement.
* Patients with uncontrolled diabetes, assessed by measuring glycosylated haemoglobin (HbA1c). (greater than to 6.4 percent )
* Potentially uncooperative patients who are not willing to go through the proposed interventions. - Moderate-to-heavy daily smokers* (who report consuming at least 11 cigarettes/day).
* Patients who are having complete lower denture
* Patients who have history of bruxism

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Crestal bone loss | 6 to 12 months
  measuring crestal bone loss around implants using periapical x ray with parallel technique in millemeters

SECONDARY OUTCOMES:
Patients satisfaction | 6 to 12 months
  Numerical Rating Scale (NRS) [11-point ordinal scale from 0 (completely dissatisfied) to 10 (completely satisfied)]